CLINICAL TRIAL: NCT01493492
Title: Urinary Proteomics Analysis for Sepsis Identification and Its Prognosis in Sepsis Patient With iTRAQ Labeling and and LC-MS/MS
Brief Title: Urinary Proteomics Analysis for Sepsis and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Other Study IDs: 20111013-007(1); 2009BAI86B03 (Other Grant/Funding Number: Chinese National Science & Technology Pillar Program)
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: SIRS; Sepsis
Keywords: proteomics,urinary,sepsis,prognosis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SIRS: 1. temperature >38 ℃ or <36℃;
  2. pulse rate>90 beats/min;
  3. ventilatory rate>20 breaths/min or hyperventilation with partial pressure of arterial carbon dioxide (PaCO2)<32mmHg;
  4. white blood cell count>12,000μL-1 or <4000μL-1 or >10% immature cells
- sepsis: Sepsis
  1. sepsis: SIRS plus infection;
  2. severe sepsis: sepsis associated with organ dysfunction, hypoperfusion, or hypotension;
  3. septic shock: sepsis with arterial hypotension, despite adequate ﬂuid resuscitation.
- non-survivors with sepsis: sepsis patients who died within 28 days

SUMMARY:
As a noninvasive examination, urinary proteomics is a very useful tool to identify renal disease. The purpose of the present study was to find differential proteins among patient with SIRS and sepsis(included survivors and non-survivors), and to screen potential biomarkers for the early diagnosis of sepsis and its prognosis. Urinary proteins were identified by iTRAQ labeling and LC-MS/MS. The bioinformatics analysis was performed with the Mascot software and the International Protein Index (IPI) and the Gene Ontology (GO) Database and KEGG pathway Database. The differentially expressed proteins were verified by Western blot by another sample collected from clinical.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years old and over;
* clinically confirmed infection;
* fulfilled at least two criteria of systemic inflammatory response syndrome
* (a) core temperature higher than 38 °C or lower than 36 °C
* (b)respiratory rate above 20/min, or PCO2 below 32 mmHg
* (c) pulse rate above 90/min, and
* (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.

Exclusion Criteria:

* younger than 18 years of age;
* acquired immunodeficiency syndrome;
* reduced polymorphonuclear granulocyte counts (< 500 μL-1);
* died within 24h after admission into the ICU, or refused to participate in the study, or declined treatment during the period of observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between May 2010 and Jan 2012 in the Respiratory ICU, Surgical ICU, and Emergency ICU, Chinese People's Liberation Army (CPLA) General Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Survival status | 28days after admited in ICU
  The survival time of patients more than 28days is defined as survival. The survival time of patients less than 28days is defined as death

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, MD, Study Director — Department of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Su L, Zhou R, Liu C, Wen B, Xiao K, Kong W, Tan F, Huang Y, Cao L, Xie L. Urinary proteomics analysis for sepsis biomarkers with iTRAQ labeling and two-dimensional liquid chromatography-tandem mass spectrometry. J Trauma Acute Care Surg. 2013 Mar;74(3):940-5. doi: 10.1097/TA.0b013e31828272c5. PMID 23425763
- [Derived] Su L, Cao L, Zhou R, Jiang Z, Xiao K, Kong W, Wang H, Deng J, Wen B, Tan F, Zhang Y, Xie L. Identification of novel biomarkers for sepsis prognosis via urinary proteomic analysis using iTRAQ labeling and 2D-LC-MS/MS. PLoS One. 2013;8(1):e54237. doi: 10.1371/journal.pone.0054237. Epub 2013 Jan 23. PMID 23372690